CLINICAL TRIAL: NCT00082511
Title: A Multi-Center, Open-Label Study to Assess the Durability and Safety of the Prevention of Bone Loss by Treatment With GL701 (Prestara™) in Women With Systemic Lupus Erythematosus Receiving Treatment With Glucocorticoids
Brief Title: GL701 (Prestara™) in Women With Systemic Lupus Erythematosus Receiving Treatment With Glucocorticoids
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Genelabs Technologies (Industry)
Responsible Party: Kenneth E. Schwartz, MD, Genelabs Technologies, Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GL03-01
Record Dates: First submitted 2004-05-11; First posted 2004-07-16 (Estimated); Last update posted 2008-01-14 (Estimated); Status verified 2008-01

CONDITIONS: Systemic Lupus Erythematosus
Keywords: Lupus; Systemic Lupus Erythematosus; SLE; Bone Loss; DHEA
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Bone Diseases, Metabolic | interventions — Dehydroepiandrosterone; GL-701

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Prasterone (GL701) — There were 4 arms to the study:
  During a previous 6 month db RCT, patients received either prasterone 200 mg/day or placebo. Upon entry into this open-label study, they were re-assigned by randomized allocation to receive either prasterone 200 mg/day or 100 mg/day. Hence, there were 4 possible treatment arms extending over the 18 months of observation between the double-blind study and the subsequent 12 month open-label extension study.

SUMMARY:
Open label safety and efficacy follow-up.

DETAILED DESCRIPTION:
This was a randomized, multi-center, open-label, parallel-group, trial of prasterone 200 or 100 mg/day for 12 months in women with lupus receiving glucocorticoid therapy who had completed an earlier 6-month randomized, placebo-controlled study (NCT00053560. Bone Mineral Density assessments were performed at baseline and at months 6 and 12.

ELIGIBILITY:
Inclusion Criteria:

* Patient has completed the full 6 month treatment period with study drug in the previous Genelabs' clinical study GL02-01.
* Concomitant treatment with prednisone (or equivalent) at a dose of ≥ 5mg/day.
* Patient has read and signed an Informed Consent Form. If the patient is not fluent in English, the Informed Consent must be signed in her native language.

Exclusion Criteria:

* Patient has had a serious study drug related adverse reaction at any time during the previous GL02-01 study.
* Any condition which in the Investigator's or Sponsor's opinion is sufficient to prevent adequate compliance with the study or likely to confuse follow-up evaluation (e.g., alcoholism, drug addiction, acute withdrawal from chemical dependency, psychiatric disease).

MEDICATIONS PROHIBITED AT ANY TIME DURING THE STUDY

* Calcitonin
* Bisphosphonates
* Fluoride at pharmacologic dose
* Strontium at pharmacologic dose
* Estrogenic steroids (except oral contraceptives)
* Selective Estrogen Receptor Modulator (raloxifene)
* Parathyroid hormone
* Any androgens, including prescription or nutritional supplement DHEA, other than study drug
* Additional Calcium supplements other than those prescribed as part of this study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2003-07; Primary Completion 2005-08 (Actual); Study Completion 2005-08 (Actual)

PRIMARY OUTCOMES:
Maintenance of bone mineral density (BMD) in women with systemic lupus erythematosus receiving glucocorticoids. | 12 months

CONTACTS AND LOCATIONS:
Locations (22):
- United States (21):
  - University of Arizona, Tucson, Arizona
  - Wallace Rheumatic Study Center, Los Angeles, California
  - Lifestyles Health Science Center, Rancho Mirage, California
  - University of California San Diego, San Diego, California
  - East Bay Rheumatology Group, San Leandro, California
  - Center for Rheumatology, Immunology and Arthritis, Fort Lauderdale, Florida
  - Rheumatology Associates of Central Florida, Orlando, Florida
  - Tampa Medical Group, P.A., Tampa, Florida
  - Northwestern University, Chicago, Illinois
  - Johns Hopkins University, Baltimore, Maryland
  - St. John's Medical Research Group, Springfield, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - SUNY Downstate Medical Center, Brooklyn, New York
  - North Shore University Hospital, Division of Rheumatology, Manhasset, New York
  - Albert Einstein Medical School, The Bronx, New York
  - Oklahoma Center for Arthritis Therapy, Tulsa, Oklahoma
  - Oregon Health & Science University, Portland, Oregon
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Sentara Medical Group DBA, Virginia Beach, Virginia
  - Seattle Rheumatology Associates, Seattle, Washington
- Immunology/Rheumatology Instituto Nacional de Ciencias Medicas y Nutricion, S.Z., Mexico City, Mexico

REFERENCES:
- [Derived] Sanchez-Guerrero J, Fragoso-Loyo HE, Neuwelt CM, Wallace DJ, Ginzler EM, Sherrer YR, McIlwain HH, Freeman PG, Aranow C, Petri MA, Deodhar AA, Blanton E, Manzi S, Kavanaugh A, Lisse JR, Ramsey-Goldman R, McKay JD, Kivitz AJ, Mease PJ, Winkler AE, Kahl LE, Lee AH, Furie RA, Strand CV, Lou L, Ahmed M, Quarles B, Schwartz KE. Effects of prasterone on bone mineral density in women with active systemic lupus erythematosus receiving chronic glucocorticoid therapy. J Rheumatol. 2008 Aug;35(8):1567-75. Epub 2008 Jul 15. PMID 18634158